CLINICAL TRIAL: NCT05093686
Title: Exploring Mechanisms of Change in a Pilot Trial of the RUBI Program in Educational Settings
Brief Title: RUBIES in Educational Settings
Acronym: RUBIES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Karen Bearss, Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCH-STUDY00003191
Record Dates: First submitted 2021-10-03; First posted 2021-10-26 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder; Disruptive Behavior
Keywords: autism; elementary schools; paraeducators; disruptive behavior
MeSH Terms: conditions — Autism Spectrum Disorder; Problem Behavior; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Simple 1:1 random assignment will be used to assign half (n=40) of the paraeducator/teacher/child triads to remote training in RUBIES, allowing for personalized delivery and tailoring of RUBIES to the paraeducator-child dyad, and the other half (n=40 dyads) to Usual Care Training (UCT, an "Autism 101" attention control condition) over a three-year period. No greater than 10% paraeducator turnover each year is expected based on prior studies.
Who Masked: Outcomes Assessor
Masking Description: Masked observers will complete the behavior observation of paraeducator use of RUBIES strategies (fidelity) and Behavior Observation of Students in School (BOSS; assessment of functional communication and classroom compliance) at all study points. Subject identity will be masked using numeric codes and only the principal investigator and research coordinator will have access to the password-protected master lists. Masked observers will receive identity coded videotapes to prevent unmasking of study condition or phase. Inclusion of UCT ensures that our behavior observation raters can remain masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RUBIES (Experimental): RUBIES provides paraeducators in training on behavioral strategies based on principles of applied behavior analysis to target student disruptive behaviors in the classroom
  Interventions: Behavioral: RUBIES
- Usual Care Treatment (Active Comparator): Usual Care Treatment provides paraeducators with foundational psychoeducation on autism spectrum disorders.
  Interventions: Behavioral: Usual Care Training

INTERVENTIONS:
Behavioral: RUBIES — RUBIES is an 8 module intervention that begins with foundational education on ASD (Session1), followed by introducing basic applied behavior analysis principles (Session 2). Instruction is then provided on strategies that can prevent problematic behaviors from occurring (Session 3 and 4). Reinforcement (Session 5) reviews the use of tangible and social reinforcers tools to promote new/desired behaviors while planned ignoring and functional communication training (Session 6) teaches that disruptive behavior can serve as a form of communication while ignoring disruptive communicative attempts. Sessions conclude with instruction on effective ways to deliver commands to promote compliance (Session 7) and targeting approaches to ensure positive behavior gains can maintain over time and strategies can be used across classrooms and staff (Session 8).
  Other Names: RUBI in Educational Settings
  Arms: RUBIES
Behavioral: Usual Care Training — Usual Care Training is an 8 module psychoeducation program that will provide foundational information on autism spectrum disorders, including the diagnostic criteria, appropriate educational services, common interventions, and how to promote social skills in the classroom.
  Arms: Usual Care Treatment

SUMMARY:
The proposed three-year pilot randomized trial aims to test the effectiveness of the newly-redesigned paraeducator-delivered RUBI for use in Educational Settings (RUBIES) intervention compared to usual care training in reducing disruptive behavior in 80 elementary-school children with ASD. Given the critical need to understand not just whether, but also how interventions work, this study also will examine paraeducator- and child-level mechanistic pathways of the RUBIES intervention.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a pervasive developmental disorder characterized by deficits in social communication and the presence of restricted and/or repetitive behavior, with prevalence estimates as high as 1 in 54 children in the US. Approximately 50% of children with ASD exhibit disruptive behaviors, such as tantrums, aggression, and noncompliance, a rate that is higher than neurotypical peers in the school environment. Disruptive behaviors impact meaningful engagement in academic tasks and with peers, as well as result in placement in more restrictive settings, higher use of restraint procedures, and suspension, all of which have lasting negative impacts. School-based behavioral management approaches, while effective, are time-consuming and resource-intensive, resulting in high costs and delays in intervention deployment. There is a need for a paradigm shift in the care model for disruptive behaviors in the classroom, specifically an efficient and pragmatic intervention model that builds capacity with direct care providers, which in turn streamlines the intervention process, reduces the need for intensive behavioral supports (thus lowering costs), and increases the number of children with ASD who can be served.

Over the past decade, the Research Units in Behavioral Interventions (RUBI) Autism Network developed and systematically tested a low-intensity (11-session) manualized intervention for parents of children ages 3 to 14 with ASD and co-occurring disruptive behavior. Results across three large scale trials have demonstrated that RUBI significantly reduces child disruptive behavior, and treatment recipients are highly engaged in the intervention. To date, no studies have evaluated the effectiveness of RUBI in schools, the most accessed service system for children with ASD.

With NIMH funding from the University of Washington ALACRITY Center grant (P50MH115837), RUBI content was iteratively redesigned in collaboration with elementary school stakeholders (administrators, teachers, paraeducators) for use in educational settings using the novel Discover, Design, Build, and Test Framework, which combines human-centered design and implementation science. In addition, target end-users (paraeducators) were identified as they: 1) provide direct support to children with ASD in both general and special education classrooms for the majority of the school day; and 2) often do not receive specialized training on effective behavioral management strategies designed to support the unique needs of children with ASD. The proposed three-year pilot randomized trial extends our work to test the effectiveness of the newly-redesigned RUBI for use in Educational Settings (RUBIES) intervention compared to usual care training (UCT) in reducing disruptive behavior in 80 elementary-school children with ASD. Given the critical need to understand not just whether, but also how interventions work, this study also will examine paraeducator- and child-level mechanistic pathways of the RUBIES intervention. Study aims include:

Aim 1: Examine the acceptability and feasibility of RUBIES with paraeducators supporting children with ASD and disruptive behavior in schools. We will measure RUBIES' acceptability (attendance, attrition, satisfaction) and feasibility (demonstration of successful study design) to determine whether paraeducators can successfully implement the RUBIES intervention in schools.

Aim 2: Conduct exploratory analyses of the impact of RUBIES compared to Usual Care Training (UCT) on disruptive behavior. Results will allow us to estimate the means, standard deviations and intraclass correlations of RUBIES compared to UCT on disruptive behavior outcomes, which will be essential for sample size/power calculations for a future definitive longitudinal RCT. Exploratory Hypothesis 1: At Week 24, children whose paraeducator was randomized to RUBIES will exhibit lower rates of observed and reported disruptive behavior compared to children whose paraeducator received UCT.

Aim 3: Conduct exploratory analyses on RUBIES' proposed paraeducator- and child-level mechanisms of change on child disruptive behavior. Exploratory Hypothesis 2: RUBIES will improve paraeducator-level mechanisms (gains in knowledge; use of more effective strategies) which will improve child disruptive behavior compared to UCT. Exploratory Hypothesis 3: RUBIES will improve child-level mechanisms (functional communication skills) which will improve child disruptive behavior compared to UCT.

Specifically, a three-year pilot effectiveness randomized controlled trial will be conducted with 80 paraeducators who support a child with ASD (n=80) from 40 public elementary schools. The child's primary teacher (N=80) and caregiver (N=80) also will be consented to contribute to outcome data on the child's behavior. Thus, 80 "triads" made up of a child-paraeducator-teacher will be enrolled. Data will be collected at baseline, Weeks 8, 12 and 24. Schools will be recruited in three cohorts that align with the school year (Years 1 and 2: N=15 schools, 30 paraeducators, 30 children with ASD, and 30 teachers; Year 3: N=10 schools, 20 paraeducators, 20 children with ASD, and 20 teachers).

Successful completion of the proposed study will allow for a large-scale effectiveness trial of RUBIES in public schools, which has the potential to improve the quality of life for children with ASD across the country.

ELIGIBILITY:
Inclusion Criteria:

* Paraeducators must be employed by the school district and work directly with children with ASD in the classroom at their school.
* Students with ASD will be included if they: 1) have a documented ASD diagnosis and a Social Responsiveness Scale-2 total raw score > 70 for males and 65 for females; 2) are enrolled in a Kindergarten-5th grade general or special education classroom and participate in a general education classroom for a minimum of 4 hours/week; 3) have a participating paraeducator; 4) have a teacher-rated Aberrant Behavior Checklist-Irritability (ABC-I) subscale score >15,; and 5) have a stable educational plan and placement.

Exclusion Criteria:

* Paraeducator is not supporting a student with autism in a general education classroom
* Student does not have a diagnosis of ASD or elevated disruptive behavior problems

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist | 24 Weeks
  After 24 weeks of treatment, students whose paraeducator received RUBIES will show greater reduction in classroom disruptive behavior as evidenced by reduction on the Aberrant Behavior Checklist Irritability Subscale compared to students whose paraeducator received Usual Care Treatment.

SECONDARY OUTCOMES:
Knowledge of Behavioral Principles | 24Weeks
  After 24 weeks of treatment, students whose paraeducator received RUBIES will show greater knowledge in behavioral principles as evidenced by higher scores on the Knowledge of Behavioral Principles measure compared to students whose paraeducator received Usual Care Treatment.
RUBIES fidelity | 24 Weeks
  After 24 weeks of treatment, paraeducators who received training in RUBIES will demonstrate observed higher implementation of evidence-based strategies based on applied behavior analysis compared to students whose paraeducator received Usual Care Treatment.
Student Behavior Observation | 24 Weeks
  After 24 weeks of treatment, students whose paraeducator received RUBIES will demonstrate lower observed rates of disruptive behavior in the classroom compared to students whose paraeducator received Usual Care Treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bearss K, Shih W, Tagavi DM, Kuo Y, Fettig A, Locke J. A Pilot Feasibility Randomized Trial of the RUBI in Educational Settings Intervention With Paraeducators Supporting Autistic Students in Public Elementary Schools. J Autism Dev Disord. 2025 Oct 15:10.1007/s10803-025-07072-8. doi: 10.1007/s10803-025-07072-8. Online ahead of print. PMID 41091357